CLINICAL TRIAL: NCT05993260
Title: Using Text Messages to Boost COVID-19 Vaccination Appointment Booking and Vaccination Rates: A Randomised Controlled Field Trial.
Brief Title: Using Text Messages to Boost COVID-19 Vaccine Booking Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Behavioural Insights Team (Other)
Collaborators: Public Health England (Other Government); Department of Health and Social Care (Unknown); NHS England (Other Government)
Responsible Party: Principal Investigator, Hannah Behrendt, Director, The Behavioural Insights Team
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021035
Record Dates: First submitted 2023-08-11; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Vaccination Hesitancy; COVID-19
MeSH Terms: conditions — Vaccination Hesitancy; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (Active Comparator): Received the text message "You are now eligible for your free NHS Covid-19 vaccine. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Control
- Simple (Experimental): Received the text message "You can now book your free NHS Covid-19 vaccine. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages
- Reserved (Experimental): Received the text message "Your free NHS Covid-19 vaccine is waiting for you. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages
- Top of queue (Experimental): Received the text message "You've reached the top of the queue and are a priority for getting a free NHS Covid-19 vaccine. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages
- Join the millions (Experimental): Received the text message "You are now eligible for your free NHS Covid-19 vaccine. Join the millions who have already had theirs. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages
- Convenience (Experimental): Received the text message "You are now eligible for your free NHS Covid-19 vaccine. Choose a time and place that suits you. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages
- Protection against virus (Experimental): Received the text message "You are now eligible for your free NHS Covid-19 vaccine. Getting vaccinated is the best protection against coronavirus. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages
- Protect you and those close to you (Experimental): Received the text message "You are now eligible for your free NHS Covid-19 vaccine. Getting the vaccine is the best way to protect yourself and those close to you against coronavirus. Please book yours now at [LINK] or by calling 119."
  Interventions: Behavioral: Behavioural science-informed text messages

INTERVENTIONS:
Behavioral: Behavioural science-informed text messages — Behaviourally-informed content in vaccination eligibility reminder text messages
  Arms: Convenience; Join the millions; Protect you and those close to you; Protection against virus; Reserved; Simple; Top of queue
Behavioral: Control — Control vaccination eligibility reminder text message
  Arms: Control

SUMMARY:
This study is a nationwide randomised controlled trial (RCT) to test the impact of behavioural science-informed text messages notifying patients of their eligibility for the COVID-19 vaccine on vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

* (i) satisfying the age criteria as defined above;
* (ii) recorded in the National Immunisation Management System (NIMS);
* (iii) with a valid mobile phone number;
* (iv) who had not already received or been invited for the COVID-19 vaccine via NIMS at the time of the study.

Exclusion Criteria:

* Participants with invalid phone numbers

Ages: 40 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1825937 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Booking rate within 72 hours | 72 hours
  The proportion of first dose vaccination appointments booked through the NHS National Booking System within 72 hours (inclusive) of the text message being sent

SECONDARY OUTCOMES:
Vaccination rate within 14 days | 14 days
  The proportion of first dose vaccinations received within 14 days (inclusive) of the text message being sent

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Behrendt, PhD, Principal Investigator — The Behavioural Insights Team
Locations (1):
- NHS England, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data requests should be submitted to NHS England and NHS Improvement (the data controller) for consideration. Access to the raw anonymised data may be granted for non-commercial research at the discretion of NHS England and NHS Improvement. Further information can be obtained from the corresponding author at hannah.behrendt@bi.team.
  Custom code that supports the findings of this study is available from the corresponding author upon request.
Supporting Information: Study Protocol, Analytic Code